CLINICAL TRIAL: NCT04126785
Title: Effects of High-Intensity Interval Versus Moderate-Intensity Continuous Heated Water-Based Exercise on Blood Pressure and Hemodynamic Variables in Older Individuals With Hypertension
Brief Title: High-Intensity Interval Versus Moderate-Intensity Continuous Water Based Exercise in Hypertensive Older Individuals
Acronym: HExOLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Emmanuel Gomes Ciolac, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECDR 1
Record Dates: First submitted 2019-09-25; First posted 2019-10-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Aging; Blood Pressure; Endothelial function; Exercise; Heart rate variability
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study 1 will be cross-over, randomized, controlled and single-blinded trial The study 2 will be randomized, parallel, controlled and single-blinded trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: In study 1 and 2 the participants will be aleatory randomized and the main investigator will perform the exercise session. The data will collected and assessed by a blinded investigator without knowledge of participants intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control without exercise in heated water-based (Placebo Comparator): CON session will perform at controlled heated water-base (30 e 32 ºC). Subject will be seated in a chair and submerged at the xiphoid process level for 30 min.
  Interventions: Other: Control Group
- High Intensity Interval Exercise in Heated Water (Experimental): High intensity interval exercise will perform at controlled heated water-base (30 e 32 ºC). Subject will be submerged at the xiphoid process level. The session will consist in 4 min walking (warm-up) at 9 level of rate perceived exertion (RPE) scale, followed by 21 min of HIIE, alternating 1 min of jogging/running at 15-17 (hard-very hard) level with 2 min of walking at 9-11 (very light-fairly light) level of RPE.
  Interventions: Other: High Intensity Interval Exercise in Heated Water-Based
- Continuous Moderate Exercise in Heated Water (Experimental): Continuous moderate exercise will perform at controlled heated water-base (30 e 32 ºC). Subject will be submerged at the xiphoid process level. The session will consist in 4 min walking (warm-up) at 9 level (light) of RPE, followed by 26 min of MICE, walking at 11-13 (fairly light) level of RPE.
  Interventions: Other: Continuous Moderate Exercise in Heated Water-Based

INTERVENTIONS:
Other: High Intensity Interval Exercise in Heated Water-Based — High intensity interval exercise will perform at controlled heated water-base (30 e 32 ºC). Subject will be submerged at the xiphoid process level. The session will consist in 4 min walking (warm-up) at 9 level of rate perceived exertion (RPE) scale, followed by 21 min of HIIE, alternating 1 min of jogging/running at 15-17 (hard-very hard) level with 2 min of walking at 9-11 (very light-fairly light) level of RPE.
  Other Names: HIIT
  Arms: High Intensity Interval Exercise in Heated Water
Other: Continuous Moderate Exercise in Heated Water-Based — Continuous moderate exercise will perform at controlled heated water-base (30 e 32 ºC). Subject will be submerged at the xiphoid process level. The session will consist in 4 min walking (warm-up) at 9 level (light) of RPE, followed by 26 min of MICE, walking at 11-13 (fairly light)level of RPE.
  Other Names: MICE
  Arms: Continuous Moderate Exercise in Heated Water
Other: Control Group — CON session will perform at controlled heated water-base (30 e 32 ºC). Subject will be seated in a chair and submerged at the until xiphoid process level for 30 min.
  Other Names: CON
  Arms: Control without exercise in heated water-based

SUMMARY:
This study will investigate the acute and chronic effects in hemodynamic and autonomic variables to high-intensity interval versus moderate-intensity continuous heated water-based exercise in older individuals with hypertension.

DETAILED DESCRIPTION:
BACKGROUND: Population aging is an unprecedented worldwide reality, which results in a change of epidemiological profile and increased prevalence of age-related non-communicable chronic diseases (NCDs). Among age-related NCDs, systemic arterial hypertension (HPT) is the leading cause of mortality and disability worldwide and has increased prevalence, morbidity and mortality with advancing age. Increase in physical activity level through regular physical exercise is one of the main global goals for the prevention and treatment of HPT and others NCDs. Among the different exercise types and intensities, high intensity interval exercise (HIIT) showed superior benefits for reducing blood pressure (BP) and improving variables involved in the pathophysiology of HPT when compared to continuous moderate-intensity exercise (MICE). However individuals with comorbidities or injures are not capable to follow adequate intensity of both types of exercise. Heated water-based has been used as an option to facilitate the individuals adherence to exercise and positive results especially in BP levels. Despite this, little is known about the effect of HIIT or MICE in heated water-based on BP and other hemodynamic variables involved in the pathophysiology of HPT in older hypertensive individuals. PURPOSE: To evaluate the hemodynamic and autonomic response to a HIIT versus MICE session and in 12 weeks of training in older individuals with hypertension. METHODS: 60 elderly hypertensives of both genders, aged over 60 years, will be randomized in the ratio 2: 2: 1 to 12 weeks of high intensity interval training (HIIT), moderate intensity continuous (MICE) or control follow-up without exercise (CON), respectively. Exercise programs will be discontinued after 12 weeks, and individuals will be followed up for another 12 weeks. Individuals will have their physical (cardiorespiratory and muscular) and functional capacity (walking, sitting and lifting ability), hemodynamic variables (blood pressure, arterial stiffness, endothelial function and cardiovascular response to exercise) and autonomic variables (variability of heart rate) and quality of life assessed before and after 12 and 24 weeks of follow-up. Before the beginning of the follow-up, 20 elderly hypertensive patients will also have a hemodynamic response (ambulatory blood pressure, endothelial function, arterial stiffness) and autonomic (heart rate variability) to a session of HI-HEx, MI-HEx and CON evaluated and compared. The feasibility of HIIE and MICE will also be assessed over the 12 weeks of its implementation. HIIT will consisted of warm up (4 min), 21 min of 1 min high intensity exercise (level 15) and "very hard" (level 17) of the subjective Rating of Perceived Exertion Scale (RPE) alternating with 2 min of walking at intensity between "easy" (level 9) and "fairly easy" (level 11) of the RPE. MICE will performed of 4 min warm up and 26 min of walking or jogging at intensity between "fairly light" (level 11) and " somewhat hard " (level 13) of the RPE.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years old;
* Hypertension diagnosed at least 6 months earlier (stage 1 or 2);
* Antihypertensive drug treatment and without dosage alteration at least 3 months earlier;
* Blood pressure inferior to 140/90 mmHg in medical office.

Non-inclusion criteria:

* Smoking individuals;
* Uncontrolled cardiovascular disease;
* Disability;
* Deficit cognitive;

Exclusion Criteria:

* Non 100% participation;
* Change (or stopped) clinical or drug treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Blood Pressure (Systolic and Diastolic) following 12 weeks of exercise. | 12 weeks
  Blood pressure will be assessed in resting (Omron HEM 7200®, Omron Healthcare Inc, Dalian, China) at the day of the sessions and using a 24 hour ambulatory blood pressure monitoring (Cardio-Mapa ®, Cardios System Ltda, Sao Paulo, Brazil), at the baseline and after 12 weeks of exercise.

SECONDARY OUTCOMES:
Effect of exercise in hemodynamic and autonomic variables assessed by endothelial function, arterial stiffness and heart rate variability | 12 weeks
  The arterial stiffness will be assessed by pulse wave velocity (Vicorder®, SMT Medical GmbH & Co., Wuerzburg, Germany) as well the endothelial function by Endocheck®. The heart rate variability will be measure using (Polar RS800CX®,Polar Electro Oy, Kempele, Finland) and 24 hour HOLTER monitoring (Cardio-Mapa ®, Cardios System Ltda, Sao Paulo, Brazil). All the measurements will be assessed at the pre and post moments of exercise protocol.
Effect of exercise in functional capacity assessed by handgrip strength test. | 12 weeks
  The handgrip strength test will assessed using Jamar®. The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles. The participant will squeeze the dynamometer with maximum isometric effort, which is maintained for about 5 seconds.The test will be performed in a single day (pre and post 12 weeks of exercise).
Effect of exercise in functional capacity assessed by 5 times sit to stand test. | 12 weeks
  The 5 times sit to stand test will measure the time taken to perform 5 repetitions of rising from a standard chair without armrest (seat height of 46 cm) to a full upright position as quickly as possible and without assistance. The test will be performed in a single day (pre and post 12 weeks of exercise), following the sequence described below, and with a 3-minute rest interval between them.
Effect of exercise in functional capacity assessed by sit and reach test. | 12 weeks
  The sit and reach test (Wells®) will be used to assess the posterior thigh and lower back flexibility. The test will be performed in a single day (pre and post 12 weeks of exercise), following the sequence described below, and with a 3-minute rest interval between them.
Effect of exercise in functional capacity assessed by timed up and go test. | 12 weeks
  The timed up and go test will be measured measured by the time to get up from a chair without armrest (seat height of 46 cm) and without assistance, walk 3 m at normal speed, turn around, walk back and sit down. The test will be performed in a single day (pre and post 12 weeks of exercise), following the sequence described below, and with a 3-minute rest interval between them.
Effect of exercise in functional capacity assessed by 6 minutes walk test. | 12 weeks
  The 6 minutes walk test will measure the distance (30 meters) that the participant can quickly walk on a flat, hard surface in a period of 6 minutes. The test will be performed in a single day (pre and post 12 weeks of exercise), following the sequence described below, and with a 3-minute rest interval between them.
Quality of Life assessed by International Physical Activity Questionnaire | 12 weeks
  The International Physical Activity Questionnaire short version (validated in the Brazilian population) will be used to assess the daily physical activity level in all volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel G Ciolac, Phd, Principal Investigator — São Paulo State University
Locations (1):
- São Paulo State Univeristy, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Participants who has interest to participated will provide an anamnesis to investigator. The investigator will analyse the IDP eligibility or not-eligibility criteria. The eligibility participant will received a document with study protocol, statistical analysis plan, informed consent form, clinical study report and analytic code informations. Thus, investigators will perform cardiopulmonary exercise test to confirm that IDP will be able to study protocol.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Initial data will be analysed at the initial sessions (cardiopulmonary exercise and functional capacity tests); at the day of sessions (study 1), after 12 weeks and 3 months of training interruption (study 2).
Access Criteria: Informed Consent Form described and signed. DP will received Informed Consent Form informing the objectives, study deling, interventions, analyses, risks and benefits. Participation in this study will be voluntary and confidential after signing of an informed consent.

REFERENCES:
- [Background] Ciolac EG, Guimaraes GV, D Avila VM, Bortolotto LA, Doria EL, Bocchi EA. Acute effects of continuous and interval aerobic exercise on 24-h ambulatory blood pressure in long-term treated hypertensive patients. Int J Cardiol. 2009 Apr 17;133(3):381-7. doi: 10.1016/j.ijcard.2008.02.005. Epub 2008 May 22. PMID 18501444
- [Background] Ciolac EG, Guimaraes GV, D'Avila VM, Bortolotto LA, Doria EL, Bocchi EA. Acute aerobic exercise reduces 24-h ambulatory blood pressure levels in long-term-treated hypertensive patients. Clinics (Sao Paulo). 2008 Dec;63(6):753-8. doi: 10.1590/s1807-59322008000600008. PMID 19060996
- [Background] Ciolac EG. High-intensity interval training and hypertension: maximizing the benefits of exercise? Am J Cardiovasc Dis. 2012;2(2):102-10. Epub 2012 May 15. PMID 22720199
- [Background] Guimaraes GV, Fernandes-Silva MM, Drager LF, de Barros Cruz LG, Castro RE, Ciolac EG, Bocchi EA. Hypotensive Effect of Heated Water-Based Exercise Persists After 12-Week Cessation of Training in Patients With Resistant Hypertension. Can J Cardiol. 2018 Dec;34(12):1641-1647. doi: 10.1016/j.cjca.2018.09.013. Epub 2018 Oct 5. PMID 30527153
- [Background] Ngomane AY, Fernandes B, Guimaraes GV, Ciolac EG. Hypotensive Effect of Heated Water-based Exercise in Older Individuals with Hypertension. Int J Sports Med. 2019 Apr;40(4):283-291. doi: 10.1055/a-0828-8017. Epub 2019 Feb 21. PMID 30791079
- [Background] Castro RE, Guimaraes GV, Da Silva JM, Bocchi EA, Ciolac EG. Postexercise Hypotension after Heart Transplant: Water- versus Land-Based Exercise. Med Sci Sports Exerc. 2016 May;48(5):804-10. doi: 10.1249/MSS.0000000000000846. PMID 26673130
- [Background] Ciolac EG, Roberts CK, da Silva JM, Guimaraes GV. Age affects exercise-induced improvements in heart rate response to exercise. Int J Sports Med. 2014 May;35(5):371-8. doi: 10.1055/s-0033-1351332. Epub 2013 Oct 15. PMID 24129990
- [Background] Ciolac EG, Carvalho VO, Guimaraes GV. High-intensity interval vs. moderate steady-state exercise. Am J Hypertens. 2010 Aug;23(8):812; author reply 813. doi: 10.1038/ajh.2010.108. No abstract available. PMID 20644524
- [Background] Ciolac EG, Bocchi EA, Bortolotto LA, Carvalho VO, Greve JM, Guimaraes GV. Effects of high-intensity aerobic interval training vs. moderate exercise on hemodynamic, metabolic and neuro-humoral abnormalities of young normotensive women at high familial risk for hypertension. Hypertens Res. 2010 Aug;33(8):836-43. doi: 10.1038/hr.2010.72. Epub 2010 May 7. PMID 20448634
- [Derived] Marcal IR, Ngomane AY, Souza FB, Ciolac EG. Hemodynamic response to heated water immersion in older individuals with hypertension. Blood Press Monit. 2021 Jun 1;26(3):171-175. doi: 10.1097/MBP.0000000000000504. PMID 33234812
- Available data/document: Brazil Research Ethics Committees: CAAE 96882818.3.0000.5398 — http://plataformabrasil.saude.gov.br/